CLINICAL TRIAL: NCT00309699
Title: Randomized, Double-Blind, Active- and Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Flexibly-Dosed Extended-Release Paliperidone Compared With Flexibly-Dosed Quetiapine and Placebo in the Treatment of Acute Manic and Mixed Episodes in Bipolar Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Flexible Doses of Extended-release (ER) Paliperidone Compared With Flexible Doses of Quetiapine and Placebo in Patients With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR010858; R076477BIM3002
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Bipolar Disorder; Mood Disorders
Keywords: Affective psychosis; mixed-state; bipolar disorder; manic disorder; manic-depressive psychosis; mania; manic state; paliperidone; paliperidone ER.
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Affective Disorders, Psychotic; Mania | interventions — Quetiapine Fumarate; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 003 (Placebo Comparator): Placebo Daily for 3 weeks
  Interventions: Drug: Placebo
- 002 (Active Comparator): Quetiapine 400 to 800 mg daily, initially titrated and flexibly dosed, for 12 weeks
  Interventions: Drug: Quetiapine
- 001 (Experimental): Paliperidone ER 3 to 12 mg daily, flexibly dosed, for 12 weeks
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Placebo — Daily for 3 weeks
  Arms: 003
Drug: Quetiapine — 400 to 800 mg daily, initially titrated and flexibly dosed, for 12 weeks
  Arms: 002
Drug: Paliperidone ER — 3 to 12 mg daily, flexibly dosed, for 12 weeks
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of flexible-doses paliperidone ER (3 to 12 mg as needed) compared with placebo over 3 weeks in patients with Bipolar I Disorder who are experiencing an acute manic or mixed episode. This study will also evaluate the effects of paliperidone ER on global functioning, and will compare the effectiveness of flexible doses of paliperidone ER to that of quetiapine over 12 weeks.

DETAILED DESCRIPTION:
Several treatments are available for the treatment of acute manic and mixed episodes associated with bipolar disorder. Some of these treatments although used for many years, are associated with well-known problems such as poor tolerability, significant toxicities, narrow therapeutic ranges, and drug interactions. Often, several drugs must be used in combination to achieve the best clinical effect. More recently, a group of compounds known as atypical antipsychotics, such as risperidone, have been licensed for use in this indication. Paliperidone has similar properties as risperidone and is expected to be as effective in the treatment of acute manic and mixed episodes associated with bipolar disorder. Paliperidone ER has been shown to be effective in schizophrenia and it has an improved drug delivery system with a reduced potential for drug interactions.

Study drug tablets are designed to deliver the appropriate amount of drug (3 mg or 6 mg) using a "Push-Pull" delivery system based on a patented oral osmotic pump technology (OROS) that allows the drug to be delivered at a relatively controlled rate for 24 hours. This study will test flexibly-dosed paliperidone ER (3 to 12 mg/day compared with placebo (inactive substance) or flexibly-dosed quetiapine (400 to 800 mg/day). There are 4 parts to the study: a screening and washout phase that lasts up to 7 days to determine if patients are eligible for the study and to discontinue all current medications, a double-blind (neither the patient nor the physician knows whether drug or placebo and what dosage is being taken) acute treatment phase that lasts for 3 weeks, a 9-week double-blind maintenance phase to see if the effects of paliperidone are maintained over a longer period, and a follow-up phase that lasts about 1 week after the final visit or early withdrawal from the study. During the acute treatment phase, patients are randomly assigned to receive treatment with placebo, 3 to 12 mg/day of paliperidone ER, or 400 to 800 mg/day of quetiapine. The dosage of paliperidone ER or quetiapine may be adjusted to meet the patient's needs. Patients who receive placebo during the acute phase (first 3 weeks) will receive paliperidone ER (beginning with 6 mg/day) during the maintenance phase (last 9 weeks). All other patients receive the same drug, i.e., either paliperidone ER or quetiapine, during both phases. The dosages during the acute phase begin at 6 mg/day for paliperidone ER and 100 mg/day for quetiapine, and may be adjusted thereafter by the study investigator to meet individual patient needs (after a forced titration of quetiapine to 400 mg/day). Patients will be hospitalized for at least the first 7 days of double-blind treatment, and may be discharged on the seventh day and followed as outpatients based on the judgment of the study doctor. End-of-study/early withdrawal procedures will be done after the last dose of study drug has been received and blood samples have been taken, or if a patient withdraws early. Patients will have a follow-up visit with safety evaluations approximately 1 week later. The study, including the screening and washout phases, will last approximately 98 days or 14 weeks.

Effectiveness will be primarily determined by the change in the total Young Mania Rating Scale (YMRS) score from the beginning (baseline) to the end of the acute treatment phase of the study. The YMRS is an 11-item established measure used to evaluate manic symptoms. A secondary measure of effectiveness is the change in the Global Assessment of Functioning (GAF) scale from baseline to the end of the acute treatment phase of the study. Other measures of effectiveness include the change from baseline to end of the maintenance phase in total YMRS score, the time to onset of therapeutic effect, responder rate (defined as 50% or more reduction from baseline in YMRS score) and changes from baseline to the end of the acute treatment phase in all other assessment scales. Additional assessment scales will be used to evaluate the clinical progress of the patient, psychotic features in bipolar disorder, quality of sleep and daytime drowsiness, health-related function, and rate the severity of the patient's bipolar disorder. Safety will be evaluated by the frequency, severity, and timing of side effects, clinical laboratory tests (including pregnancy tests), 12-lead electrocardiograms (ECGs), vital signs measurements, and physical and neurological examinations.

The study hypotheses for the primary and secondary effectiveness measures are that 1) flexibly dosed (dosages of 3 to 12 mg/day) paliperidone ER have more effect than placebo on the change from baseline in the YMRS total score at the end of 3 weeks of treatment, 2) flexibly-dosed paliperidone ER has more effect than placebo on the change from baseline in GAF score at the end of 3 weeks of treatment, and 3), flexibly-dosed paliperidone ER is not worse than quetiapine in the change in YMRS score at 12 weeks. The potential effect on the variation in genes related to paliperidone ER may be evaluated separately in patients who consent to DNA (deoxyribonucleic acid) testing. All study drug will be administered twice daily. The dosages during the acute phase (first 3 weeks) begin at 6 mg/day for paliperidone ER and 400 mg/day for quetiapine (after a forced titration from 100 mg/day), and may be adjusted thereafter by the investigator to meet individual patient needs within the ranges of 3-12 mg/day and 400-800 mg/day. Patients who receive placebo during the acute phase will receive paliperidone ER (starting with 6 mg/day) during the maintenance phase (last 9 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM IV) criteria for Bipolar I Disorder, Most Recent Episode Manic or Mixed (with or without psychotic features)
* history of at least 1 previously documented manic or mixed episode requiring medical treatment within 3 years before the screening phase
* total score of at least 20 on the YMRS at screening and at baseline
* if taking mood stabilizers, antipsychotics, or antimanic drugs, must have discontinued that medication at least 3 days before baseline
* women must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or agree to practice an effective method of birth control if they are sexually active before entry and throughout the study (effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier method, and male partner sterilization)
* able and willing to comply with self-administration of medication, or have consistent help or support available.

Exclusion Criteria:

* Meets DSM-IV criteria for rapid cycling and schizoaffective disorder
* In the opinion of the study doctor, is at significant risk for suicidal or violent behavior during the course of the study
* Has used cocaine, phencyclidine, amphetamine, methylphenidate, pemoline, an opioid (excluding codeine), hallucinogen, or any other drug that may be associated with manic symptoms as evidenced by a positive urine drug screen
* Has received benzodiazepines at doses equal to 4 mg/day of lorazepam or higher for a period of 3 months or longer immediately before the screening phase.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2006-04; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness outcome is the change in the total YMRS score from baseline to the last assessment during the acute treatment phase. | 3 weeks

SECONDARY OUTCOMES:
The secondary effectiveness outcomes are the change in GAF from baseline to endpoint or the last assessment during the acute treatment phase and the change in total YMRS score from baseline to endpoint or the last assessment during the maintenance phase. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (47):
- United States (22):
  - Cerritos, California
  - Garden Grove, California
  - Oceanside, California
  - San Diego, California
  - Bradenton, Florida
  - Fort Lauderdale, Florida
  - Kissimmee, Florida
  - Maitland, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Prairie Village, Kansas
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Flowood, Mississippi
  - Clementon, New Jersey
  - Moore, Oklahoma
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Dallas, Texas
- Athens, Greece
- Lithuania (2):
  - Alytus
  - Vilnius
- Russia (7):
  - Kazan'
  - Lipetsk
  - Moscow Region
  - Moscow Russia
  - Nizny Novgorod
  - Saratov
  - St-Petersburg Na
- South Korea (2):
  - Incheon
  - Seoul
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Taichung
  - Taipei
- Turkey (Türkiye) (3):
  - Ankara
  - Diyarbakır
  - Istanbul
- Ukraine (6):
  - Donetsk
  - Hlevakha
  - Kharkiv
  - Kiev
  - Odesa
  - Simferopol

REFERENCES:
- [Derived] Vieta E, Nuamah IF, Lim P, Yuen EC, Palumbo JM, Hough DW, Berwaerts J. A randomized, placebo- and active-controlled study of paliperidone extended release for the treatment of acute manic and mixed episodes of bipolar I disorder. Bipolar Disord. 2010 May;12(3):230-43. doi: 10.1111/j.1399-5618.2010.00815.x. PMID 20565430
- See also: A Study to Evaluate the Efficacy and Safety of Flexible Doses of Extended-Release (ER) Paliperidone Compared With Flexible Doses of Quetiapine and Placebo in Patients With Bipolar I Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=722&filename=CR010858_CSR.pdf